CLINICAL TRIAL: NCT02783911
Title: Comparison of Clinical and Radiographic Success Between Mineral Trioxide Aggregate (MTA) & Ferric Sulfate (FS) Pulpotomies for Primary Molars
Brief Title: Comparison of Mineral Trioxide Aggregate (MTA) & Ferric Sulfate (FS) Pulpotomies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The resident graduated.
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Jung-Wei Chen, DDS, MS, PhD, Pediatric Dental Director, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5140262
Record Dates: First submitted 2016-05-18; First posted 2016-05-26 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Primary Teeth; Pulpotomy
Keywords: Clinical and Radiograph
MeSH Terms: interventions — ferric sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mineral Trioxide Aggregate (Experimental): Subject with pulpotomy treated with MTA MTA paste (< 1gm) will be placed on pulp orifice once for the life of the primary teeth
  Interventions: Device: MTA
- Ferric Sulfate (Experimental): Subject with pulpotomy treated with FS FS paste (<1gm) will placed on pulp orifice once for 15 secs and removed on primary teeth
  Interventions: Drug: Ferric Sulfate

INTERVENTIONS:
Device: MTA — Mineral Trioxide Aggregate grey paste
  Arms: Mineral Trioxide Aggregate
Drug: Ferric Sulfate — Ferric Sulfate paste
  Other Names: FS
  Arms: Ferric Sulfate

SUMMARY:
Comparison of clinical and radiographic success between Mineral Trioxide Aggregate and Ferric Sulfate pulpotomies for primary molars. Recall appointments are completed 6 months, 9 months and 12 months.

DETAILED DESCRIPTION:
Comparison of clinical and radiographic success between Mineral Trioxide Aggregate and Ferric Sulfate pulpotomies for primary molars. Recall appointments are completed 6 months, 9 months and 12 months. Regular recall and follow up will be performed for patients who has MTA or FS pulpotomies. Clinical and radiographic findings will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II
* Primary Molars diagnosed with normal or reversible pulpitis with vital carious pulp exposures
* Teeth that can have hemostasis can be achieved with pressure
* No clinical symptoms
* No radiographic signs of internal resorption or external root resorption

Exclusion Criteria:

* Primary Molars diagnosed with irreversible pulpitis or necrotic pulp
* Teeth that can not achieve hemostasis
* Teeth with abscess or fistula
* Teeth that have radiographic signs of internal resorption or external resorption

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Wei Chen, DDS,MS,PhD, Principal Investigator — Loma Linda University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asgary S, Shirvani A, Fazlyab M. MTA and ferric sulfate in pulpotomy outcomes of primary molars: a systematic review and meta-analysis. J Clin Pediatr Dent. 2014 Fall;39(1):1-8. doi: 10.17796/jcpd.39.1.b454r616m2582373. PMID 25631717
- [Result] Yildirim C, Basak F, Akgun OM, Polat GG, Altun C. Clinical and Radiographic Evaluation of the Effectiveness of Formocresol, Mineral Trioxide Aggregate, Portland Cement, and Enamel Matrix Derivative in Primary Teeth Pulpotomies: A Two Year Follow-Up. J Clin Pediatr Dent. 2016 Winter;40(1):14-20. doi: 10.17796/1053-4628-40.1.14. PMID 26696101
- [Result] Stringhini Junior E, Vitcel ME, Oliveira LB. Evidence of pulpotomy in primary teeth comparing MTA, calcium hydroxide, ferric sulphate, and electrosurgery with formocresol. Eur Arch Paediatr Dent. 2015 Aug;16(4):303-12. doi: 10.1007/s40368-015-0174-z. Epub 2015 Apr 2. PMID 25833280
- [Result] Frenkel G, Kaufman A, Ashkenazi M. Clinical and radiographic outcomes of pulpotomized primary molars treated with white or gray mineral trioxide aggregate and ferric sulfate--long-term follow-up. J Clin Pediatr Dent. 2012 Winter;37(2):137-41. doi: 10.17796/jcpd.37.2.j3h27p624u163868. PMID 23534318

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3-10 years old, deep caries, No radiographic signs of internal/external root resorption, No pathology change, no swelling or abscess.
Units Other Than Participants: tooth
Period: Overall Study
Arm/Group | Mineral Trioxide Aggregate | Ferric Sulfate
Started | 11; 12 tooth | 46; 53 tooth
Completed | 8; 9 tooth | 14; 15 tooth
Not Completed | 3; 3 tooth | 32; 38 tooth
Not completed — Lost to Follow-up | 3 | 32

BASELINE CHARACTERISTICS:
Population: some participants has more than one tooth needs pulpotomy treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Mineral Trioxide Aggregate | Ferric Sulfate | Total
Number analyzed (Participants) | 11 | 46 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 46 | 57
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 73.9 (16.9) | 81.3 (19.9) | 78.5 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 3 | 29 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
patient has deep caries [Count of Participants; unit: Participants] | 11 | 46 | 57

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Clinical Success Between Mineral Trioxide Aggregate (MTA) & Ferric Sulfate (FS) Pulpotomies in Primary Molars
Description: At recall visits 6,9,12 months, blinded clinical examination will be completed by participating faculty members who are calibrated to clinical scaring criteria. Periapical radiographs will be taken and evaluated by 2 pediatric dentists and 1 endodontist, for presence of various pathologies. Scored based on the criteria established by Zurn and Seale 2008. Scores will be transferred to Microsoft Excel. The difference between the two materials will be analyzed using the Mann-Whiteney U test, chi-square test and Fisher's exact test. Intra- and inter-rater agreement will be measured for radiographic assessment using Cohen's kappa test
Time Frame: 1 year
Population: The patients who came back for follow up for long term clinical and radiographic success.
Measure: Count of Units; unit: tooth
Units Other Than Participants: tooth
Arm/Group | Mineral Trioxide Aggregate | Ferric Sulfate
Number analyzed (Participants) | 8 | 14
Number analyzed (tooth) | 9 | 15
tooth
  Clinical success | 7 | 11
  Clinical fail | 2 | 4
Statistical Analysis 1: Comparison: Mineral Trioxide Aggregate vs Ferric Sulfate; Test type: Superiority; p = 0.808, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Mineral Trioxide Aggregate | Ferric Sulfate
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/46
Other Adverse Events (participants affected / at risk) | 0/11 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT02783911/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT02783911/SAP_001.pdf
  • Informed Consent Form (2015-01-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT02783911/ICF_002.pdf